CLINICAL TRIAL: NCT03836794
Title: Does Geography and Place of Residence Affect Cancer Care: An Interview Study
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-109-18
Record Dates: First submitted 2019-01-24; First posted 2019-02-11 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is existing evidence that rural cancer patients tend to have worse survival outcomes. Potential reasons include: differences in endurance of coping with illness, different attitudes about illness, the nature of rural lifestyles, and poorer access to healthcare services. Some of these factors may affect their delay in presentation of cancer, and/or delay in seeking treatment in a timely manner. Differences in health outcomes between urban and rural populations have been described in a number of health conditions, and to date survival/health outcomes related to cancer have been the most extensively researched. Rurality has been associated with negative impacts on cancer outcomes in studies from the United Kingdom and elsewhere. However, as with rural health disadvantage overall, the underlying causes are uncertain. There is some evidence that rural populations are less likely to engage with screening services and receive lower rates of chemotherapy and surgery. If restricted access to services was the major determinant of poorer cancer outcomes for rural populations, this should also be reflected in longer delays to diagnosis and treatment for cancer for those patients living more remotely. However, a recent study from the Northeast of Scotland contradicts this, finding that rural patients in Scotland were diagnosed and treated for their cancers quicker than their urban counterparts, but died earlier . The investigator's proposed research aims to provide insights into differences between how urban and rural patients engage with health services in National Health Service (NHS) Grampian by interviewing patients about their diagnostic pathway, their interactions with the healthcare service, their treatment choices, and how these may have been influenced by where they live.

DETAILED DESCRIPTION:
A review of literature and data analysis within the Northeast Aberdeen Scotland Cancer and Residence (NASCAR) database has established that although rural patients are diagnosed and treated much more quickly than their urban counterparts, they are significantly more likely to die in the first year after diagnosis. At times, it was found that patients voluntarily opted out of certain recommended regimens such as radiotherapy simply due to the burden of travel. Currently, literature only proposes themes such as stoicism, attitudes, the nature of rural lifestyles, and access to healthcare services, but nothing is explicitly defined. Rural living may influence healthcare interaction at multiple levels and the potentially complex effect on cancer outcomes is best addressed through qualitative research with both urban and rural patients. Qualitative enquiries are most likely to give insights into potential mechanisms of urban/rural inequality within Northeast Scotland beyond.

The Social Ecological Model (SEM) is a theory-based framework for understanding the multifaceted and interactive effects of personal and environmental factors that determine behaviours, and for identifying behavioural and organisational leverage points and intermediaries for health promotion within organisations (9). This model includes several nested levels; individual, interpersonal, community, organisational, and policy. When addressing any health issue, it is important to assess how every level influences one another. In our systematic literature review, the investigators found that the SEM provided an explanatory framework through which to explore potential inequalities in urban and rural cancer outcomes. Within interviews, the investigators will use the theoretical framework to prompt participants.

Phase 1: Identifying eligible patients and recruitment Patients will be recruited from two sources. First, those from rural areas and residing at the CLAN House residence Westburn Road, Aberdeen during an episode of hospital-based cancer care will be approached by CLAN staff on behalf of the researchers. Second, patients attending oncology clinic D at Aberdeen Royal Infirmary will be approached by clinic staff on behalf of researchers. Interested patients will be directed to the researcher provided the Patient Information Sheet from Clan/ARI staff to obtain more information about the study and be invited to complete the consent process.

Phase 2: Interviews with consented cancer patients. Consenting research participants will be interviewed on a single occasion by Miss Carriere, using a semi-structured approach. Interviews will be digitally audio recorded with permission from the participant. The interview will take approximately 45 minutes. The interview will happen at a place of the participant's own choosing such as within the University of Aberdeen, Clinic D - Aberdeen Royal Infirmary (ARI), or CLAN locations. There will also be an option to conduct telephone interviews which will last approximately 45 minutes.

Phase 3: Transcribing data from interviews and coding them appropriately Miss Carriere or NJC Secretarial, who is a member of university staff in Academic Primary Care will transcribe all interviews after they occur and which is an approved third party organisation for transcribing such work. Miss Carriere will also utilise a 'Contact Sheet' to record impressions of the participant not picked up by audio-recorded data (Miles and Huberman). This will take up to 6 months to complete and analyse. Participant interviews will be transcribed verbatim for analysis. Framework analysis using components of the socio-ecological model, a coding framework of the main themes and sub themes will be established (9). NVivo version 12 software will be used to assist with the management of the data. A sample of manuscripts will be coded by a second researcher to ensure validity.

Phase 4: Disseminate information gathered from interviews Study results will be collated in the form of a manuscript and further expanded in a PhD thesis. At the time of the interview, participants will be asked to if they would like to receive a copy of their manuscript. Before publication of the manuscript, any participants requesting to be kept informed of results will be emailed a copy of the final study report or a lay summary of the results will be published and available.

Data Management Digital audio-recordings will be transcribed by Miss Carriere or transcribed by NJC Secretarial and all data will be anonymised by Miss Carriere according to unique participant identification codes. NJC Secretarial will receive a copy of the audio recorded files with only the anonymous study ID number via secure file transfer service ZendTo hosted by University of Aberdeen. NJC Secretarial will transcribe this data, sending the transcription back to Romi Carriere via Zend to. Audio recordings would then be deleted by NJC Secretarial. Transcripts will be imported into NVivo version 12, and each participant will be assigned a Study ID that will de-identify their private information. This study ID will be stored separately from the other data and will only be accessed by the research team. Data will be securely stored within and excel file within a secure server and/or locked cabinet in the Institute of Applied Health Sciences at the University of Aberdeen. All study documentation will be kept for at least 10 years after publication of the study data in accordance with the sponsors archiving Standard Operating Procedure (SOP).

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible to participate if they are adults, 18 years or over, confirmed cancer diagnosis from the top eight cancer sites (lung, oesophageal, colorectal, breast, pancreatic, prostate, kidney, and bladder) within the last 2 years. Participants can have all stages and all grades of cancer as long as they feel able to provide a full interview for approximately 45 minutes. There will be an opportunity for patient to opt into telephone interviews. Interviewees are able to stop their interviews at any moment without having to give a reason.

Exclusion Criteria:

* The research team involved in recruiting will exclude patients that are unable to give consent, non-English speaking patients, patients under the age of 18 and patients that are too ill based on the observation of the clinical staff.

This study will exclude persons who have difficulty understanding verbal explanations in English. This study is a small qualitative study based upon interviews conducted by a single researcher in the English language. The analysis of the data will depend upon specific words and utterances which are used by the participant. Meaning will be derived from words, phrases, and utterances and will be reliant upon the participant being able to communicate in the English language.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The recruited population will be newly diagnosed cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Qualitive Measures of a Study Questionnaire | 1 year
  Interviewing 25 patients, rich, explanatory qualitative data from patients about their path to diagnosis and their path to treatment and how that may have been influenced by where they live.

CONTACTS AND LOCATIONS:
Overall Officials: Romi A Carriere, MPH, Principal Investigator — University of Aberdeen
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonelli M, Wiebe N, Fortin M, Guthrie B, Hemmelgarn BR, James MT, Klarenbach SW, Lewanczuk R, Manns BJ, Ronksley P, Sargious P, Straus S, Quan H; Alberta Kidney Disease Network. Methods for identifying 30 chronic conditions: application to administrative data. BMC Med Inform Decis Mak. 2015 Apr 17;15:31. doi: 10.1186/s12911-015-0155-5. PMID 25886580
- [Background] Carriere R, Adam R, Fielding S, Barlas R, Ong Y, Murchie P. Rural dwellers are less likely to survive cancer - An international review and meta-analysis. Health Place. 2018 Sep;53:219-227. doi: 10.1016/j.healthplace.2018.08.010. Epub 2018 Sep 5. PMID 30193178
- [Background] Jones AP, Haynes R, Sauerzapf V, Crawford SM, Zhao H, Forman D. Travel time to hospital and treatment for breast, colon, rectum, lung, ovary and prostate cancer. Eur J Cancer. 2008 May;44(7):992-9. doi: 10.1016/j.ejca.2008.02.001. Epub 2008 Mar 28. PMID 18375117
- [Background] Campbell NC, Elliott AM, Sharp L, Ritchie LD, Cassidy J, Little J. Impact of deprivation and rural residence on treatment of colorectal and lung cancer. Br J Cancer. 2002 Sep 9;87(6):585-90. doi: 10.1038/sj.bjc.6600515. PMID 12237766
- [Background] Jones AP, Haynes R, Sauerzapf V, Crawford SM, Zhao H, Forman D. Travel times to health care and survival from cancers in Northern England. Eur J Cancer. 2008 Jan;44(2):269-74. doi: 10.1016/j.ejca.2007.07.028. Epub 2007 Sep 20. PMID 17888651
- [Background] Lin CC, Bruinooge SS, Kirkwood MK, Olsen C, Jemal A, Bajorin D, Giordano SH, Goldstein M, Guadagnolo BA, Kosty M, Hopkins S, Yu JB, Arnone A, Hanley A, Stevens S, Hershman DL. Association Between Geographic Access to Cancer Care, Insurance, and Receipt of Chemotherapy: Geographic Distribution of Oncologists and Travel Distance. J Clin Oncol. 2015 Oct 1;33(28):3177-85. doi: 10.1200/JCO.2015.61.1558. Epub 2015 Aug 24. PMID 26304878
- [Background] Turner M, Fielding S, Ong Y, Dibben C, Feng Z, Brewster DH, Black C, Lee A, Murchie P. A cancer geography paradox? Poorer cancer outcomes with longer travelling times to healthcare facilities despite prompter diagnosis and treatment: a data-linkage study. Br J Cancer. 2017 Jul 25;117(3):439-449. doi: 10.1038/bjc.2017.180. Epub 2017 Jun 22. PMID 28641316
- [Background] Williams S, Bi P, Newbury J, Robinson G, Pisaniello D, Saniotis A, Hansen A. Extreme heat and health: perspectives from health service providers in rural and remote communities in South Australia. Int J Environ Res Public Health. 2013 Oct 29;10(11):5565-83. doi: 10.3390/ijerph10115565. PMID 24173140
- [Background] Murage P, Murchie P, Bachmann M, Crawford M, Jones A. Impact of travel time and rurality on presentation and outcomes of symptomatic colorectal cancer: a cross-sectional cohort study in primary care. Br J Gen Pract. 2017 Jul;67(660):e460-e466. doi: 10.3399/bjgp17X691349. Epub 2017 Jun 5. PMID 28583943